CLINICAL TRIAL: NCT04525209
Title: Integrative Proteomic Characterization of Pancreatic Ductal Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, HAOCHEN, Chen Hao, Ruijin Hospital
Other Study IDs: 2020-08-20
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Tumor Tissues and Non-tumor Tissues From PDAC Patients Were Used for Genomic and Transcriptome Sequencing Analysis and Proteomics and Phosphorylated Proteomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PDAC tumor and Non-tumor DNA, RNA, protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A large-scale, high-throughput, multi-dimensional comprehensive study of PDAC multiomics will be carried out. In this study, clinical specimens of resected PDAC collected by our research group from 2017 to 2019 will be selected as research objects.Tumor tissues and their adjacent non-tumor tissues from more than 200 PDAC patients are expected to be used for genome, transcriptome sequencing and mass spectrometry analysis of proteome and phosphorylated proteome.Combined with the data results of multiomics, bioinformatics analysis and network database information, we will clarify the relationship between multiomics of pancreatic cancer and established the new subtyping of pancreatic cancer proteome. A molecular landscape of the progression of pancreatic cancer at the genome-transcriptome-proteome level provides new therapeutic targets to improve the prognosis of this deadly disease.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of pancreatic cancer was confirmed by histological examination or fine needle aspiration cytology;
2. The tumor was graded according to THE WHO standard, and the tumor stage was graded according to the TNM stage;

Exclusion Criteria:

1. The inclusion criteria of the above groups were not met;
2. There are few tissue specimens, only enough for clinical diagnosis;
3. Patients are unwilling to conduct follow-up study;
4. For the new diagnosed patient, radiotherapy or chemotherapy have been given in the previous three months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese PDAC patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Integrative Proteomic Characterization of PDAC | Two yeaers
  The genome-transcriptome proteome level provides a molecular landscape of the progression of pancreatic cancer, providing new therapeutic targets to improve the prognosis of PDAC

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- RUIJIN Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao Q, Zhu H, Dong L, Shi W, Chen R, Song Z, Huang C, Li J, Dong X, Zhou Y, Liu Q, Ma L, Wang X, Zhou J, Liu Y, Boja E, Robles AI, Ma W, Wang P, Li Y, Ding L, Wen B, Zhang B, Rodriguez H, Gao D, Zhou H, Fan J. Integrated Proteogenomic Characterization of HBV-Related Hepatocellular Carcinoma. Cell. 2019 Oct 3;179(2):561-577.e22. doi: 10.1016/j.cell.2019.08.052. PMID 31585088
- [Result] Cancer Genome Atlas Research Network. Electronic address: andrew_aguirre@dfci.harvard.edu; Cancer Genome Atlas Research Network. Integrated Genomic Characterization of Pancreatic Ductal Adenocarcinoma. Cancer Cell. 2017 Aug 14;32(2):185-203.e13. doi: 10.1016/j.ccell.2017.07.007. PMID 28810144